CLINICAL TRIAL: NCT03558581
Title: Nursing Interventions for Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Elizabeth Prado Lima Figueiredo, Associate Professor, Pontificia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EnfDiaTrial
Record Dates: First submitted 2018-04-30; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus; Chronic Kidney Diseases
Keywords: Nursing Process; Nephrology Nursing; Education Health
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients have not received any special intervention, the follow up care was the standard care for the specific clinic
- Intervention (Experimental): After initial allocation the select patient received six educational interventions selected from Nursing Intervention Classification (NIC)
  Interventions: Other: Educational

INTERVENTIONS:
Other: Educational
  Other Names: Teaching: individual and Teaching: disease process.; Control of hyperglycemia and Control of hypoglycemia.; Teaching: prescription drugs; Teaching: psychomotor skills.; Teaching: Foot care.; Teaching: activity / prescribed exercises.
  Arms: Intervention

SUMMARY:
Introduction: Diabetes mellitus (DM) is a very frequent pathology, which can lead to renal failure and the need for renal replacement therapy. In people with chronic kidney disease (CKD) and diabetes mellitus (DM), glycemic control is very important for the prevention of microvascular injury. In this context, the Nursing Process (NP) is the instrument to guide care, contributing to the attention of individuals' needs. Objective: To evaluate the results of Nursing Outcomes Classification (NOC), obtained through interventions of the Nursing Interventions Classification (NIC) for the glycemic control, in patients with diabetes in renal replacement therapy, with a diagnosis of Unstable Glycemia, of the North American Nursing Diagnosis - International (NANDA-I). Method: Randomized clinical trial in three dialysis services in southern Brazil. Population: Type I and II diabetes patients on hemodialysis. Sample: Over 18 years old, literate, who accept to participate in the study by signing a Term of Consent Free and Clarified. Exclusion criteria: severe uncorrected deficiency in hearing, speech, total amaurosis, degenerative neurological diseases, or score less than 20 in the Mini Mental State Examination. Randomization occurred by clusters, considering dialysis shifts. The CG followed routine treatment and guidelines, while the IG received nursing interventions on a monthly basis for 6 months. Variables related to NOC scores and the knowledge, attitude and self-care tests for DM were applied before and after the intervention period. After the intervention period, a washout period of 06 months will occur, after which the variables will be collected.

DETAILED DESCRIPTION:
After randomization, the intervention group was assesses by a nurse determining the nursing outcomes (NOC)for the specific nursing diagnosis Unstable glycemia. One educational intervention per month was done:

1. Teaching: individual and Teaching: disease process.
2. Control of hyperglycemia and Control of hypoglycemia.
3. Teaching: prescription drugs (prescription drugs, was carried out focusing on oral hypoglycemic agents and insulin)
4. Teaching: psychomotor skills ( was performed with a view to the management and application of insulin). In case of use oral antiglycemic agent the Teaching: prescription drugs and control of hyperglycaemia and hypoglycemia was repeated
5. Teaching: Foot care.
6. Teaching: activity / prescribed exercises. After the completion of the six intervention patients were assessed for outcome classification the study will contemplate a 6 months washout between the NOC assessment ( end of interventions and final assessment)

ELIGIBILITY:
Inclusion Criteria:

* diabetic with chronic kidney disease on hemodialysis
* over 18 years old
* literate,
* who accept to participate in the study by signing a Term of Consent Free and Clarified

Exclusion Criteria:

* severe uncorrected deficiency in hearing, speech,
* total amaurosis,
* degenerative neurological diseases,
* score less than 20 in the Mini Mental State Examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Glycemic control - HbA1< 7% | 1 year
  blood sample after NIC interventions

SECONDARY OUTCOMES:
Improve Knowledge assessed by questionaries DKNA | 1 year
  DKNA has 15 multiple choice response items and covers aspects related to the general knowledge of diabetes mellitus. The questions are about basic physiology, food groups and substitutions, DM management in case of complications, and general principles of disease care).
  The measurement scale used is from 0 to 15. A score (1) is assigned for correct answer and zero (0) for incorrect. Score greater than eight indicates knowledge about diabetes mellitus

OTHER OUTCOMES:
Improve attitude and coping of Diabetes assessed by questionaries ATT-19 | 1 year
  ATT - 19, it is an instrument that seeks the psychological adjustment measure for diabetes mellitus, developed as a response to the needs of evaluation of psychological and emotional aspects of the disease. It contains nineteen items that include six factors: a) stress associated with DM, b) receptivity to treatment, c) trust in treatment, d) personal efficacy, e) health perception, f) social acceptance, whose responses are measured through five-point Likert scale (I totally disagree - score 1, until I fully agree - score 5). The total value of the score varies from from 19 to 95 points. A score greater than 70 points indicates a positive attitude about the disease

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Capellari, Master, Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul; Ana Figueiredo, PhD, Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul
Locations (1):
- Pontificia Universidade Católica Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No